CLINICAL TRIAL: NCT06591468
Title: A Multicenter, Randomized, Controlled Trial of Prednisone Combined With Ursodeoxycholic Acid in the Treatment of Primary Biliary Cholangitis With Moderate to Severe Interface Hepatitis Characteristics
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Ying (Other)
Responsible Party: Sponsor-Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242283
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-06

CONDITIONS: Primary Biliary Cholangitis (PBC)
Keywords: Primary Biliary Cholangitis; interface hepatitis; Ursodeoxycholic Acid; Corticosteroids
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Prednisone; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone (Experimental): Combination therapy of UDCA (13-15 mg/kg/day) and prednisone. Prednisone 30-40 mg/day, at 7am in the morning, gradually reduced after 1 month (5mg every 7-14 days) to 5-10 mg for maintenance treatment
- UDCA (Active Comparator): UDCA (13-15 mg/kg/day)
  Interventions: Drug: UDCA (Ursodeoxycholic acid)

INTERVENTIONS:
Drug: Prednisone — Prednisone 30-40 mg/day, at 7am in the morning, gradually reduced after 1 month (5mg every 7-14 days) to 5-10 mg for maintenance treatment
Drug: UDCA (Ursodeoxycholic acid) — 13-15 mg/kg/day
  Arms: UDCA

SUMMARY:
About 1/3 of patients with primary biliary cholangitis (PBC) exhibit moderate to severe interface hepatitis, and this group of patients have poor response to UDCA treatment. However, as it is not yet sufficient to diagnose autoimmune hepatitis or overlap syndrome, it is difficult to initiate immunosuppressive therapy such as steroids according to current guidelines. The aim of this study is to explore whether PBC patients with moderate to severe interfacial inflammation can benefit from UDCA combined with prednisone therapy, and its treatment safety.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily joining the group, able to understand and sign an informed consent form;
2. 18 years old ≤ age ≤ 75 years old;
3. The diagnosis of primary biliary cholangitis follows the AASLD international diagnostic and treatment guidelines (meeting two of the following three criteria: AMA or gp210, sp100 positive; Elevated serum ALP levels; Pathological manifestations include non suppurative cholangitis and destruction of the interlobular bile duct;
4. Liver histology suggests moderate to severe interfacial hepatitis (moderate,<50% portal or fibrous septa destruction, severe,>50% portal or fibrous septa destruction) with serum ALT<5 * ULN, serum IgG<2 * ULN, and negative serum anti smooth muscle antibodies;
5. Not receiving UDCA, hormone or other immunosuppressive therapy before enrollment;
6. ALP>1.67 * ULN.

Exclusion Criteria:

* History or presence of other concomitant liver diseases.
* ALT or AST > 5×ULN, TBIL > 3×ULN.
* If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.
* Allergic to fenofibrate or ursodeoxycholic acid.
* Taking hepatotoxic drugs (e.g., dapsone, erythromycin, fluconazole, ketoconazole, rifampicin) for more than 2 weeks within 6 months, and long-term hormonal users.
* Recurrent variceal bleeding, poorly controlled hepatic encephalopathy or refractory ascites.
* Patients with a history of severe cardiac, cerebrovascular, renal, respiratory disease or functional failure, and psychiatric disorders (including those due to alcohol and drug abuse).
* Creatinine >1.5×ULN and creatinine clearance <60 ml/min.
* Currently using statins (such as pravastatin, fluvastatin, and simvastatin), other fibrates (such as gemfibrozil and bezafibrate), and drugs structurally similar to fenofibrate (like ketoprofen).
* Planned to receive an organ transplant or an organ transplant recipient.
* Needing Liver transplantation within 1 year according to the Mayo Rick score.
* Any other condition(s) that would compromise the safety of the subject or compromise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with biochemical response | 1 year
  Alkaline Phosphatase < 1.67*ULN

SECONDARY OUTCOMES:
Assessment of the pruritus and fatigue | 1, 3, 6, 9, and 12 months
  Change From Baseline in Fatigue and Pruritus as Assessed by Visual Analogue Scale (VAS) Total Score for Fatigue and Pruritus. (0-10, higher scires mean a worse outcome)
Survival without transplantation and hepatic impairment | 1 year
  Occurrence of ascites, variceal bleeding, hepatic encephalopathy, liver-transplantation, or death.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Xijing hospital, Xi'an, Shaanxi